CLINICAL TRIAL: NCT01336088
Title: Phase 2, Randomized, Double-blind, Placebo-controlled, Parallel Group, Multicenter Study to Evaluate the Safety, Tolerability and Efficacy of ADX48621 in the Treatment of Levodopa Induced Dyskinesia in Patients With Parkinson's Disease
Brief Title: ADX48621 for the Treatment of Levodopa Induced Dyskinesia in Patients With Parkinson's Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Addex Pharma S.A. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ADX48621-201
Record Dates: First submitted 2011-04-04; First posted 2011-04-15 (Estimated); Last update posted 2012-07-16 (Estimated); Status verified 2012-07

CONDITIONS: Parkinson's Disease
Keywords: dyskinesia; Parkinson's disease
MeSH Terms: conditions — Parkinson Disease; Dyskinesias | interventions — 6-fluoro-2-(4-(pyridin-2-yl)but-3-yn-1-yl)imidazo(1,2-a)pyridine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- ADX48621 (Experimental)
  Interventions: Drug: ADX48621
- ADX48621 Matching Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: ADX48621 — oral administration
  Other Names: Dipraglurant
  Arms: ADX48621
Drug: Placebo — oral administration
  Arms: ADX48621 Matching Placebo

SUMMARY:
The primary objective of the study is to evaluate the safety and tolerability of ADX48621 in Parkinson's disease patients following four weeks of dosing.

The secondary objectives of the study include the evaluation of the efficacy of ADX48621 compared with placebo in reducing levodopa induced dyskinesia in patients with Parkinson's; the evaluation of the effect of ADX48621 on symptoms of Parkinson's disease and patient ability to function, and the evaluation of the effect of coadministration of ADX48621 on L-dopa efficacy.

DETAILED DESCRIPTION:
First study of ADX48621 in male and female Parkinson's disease patients with levodopa-induced dyskinesia. Four weeks, double-blind, placebo-controlled dose titration from 50 mg once daily up to 100 mg three times daily, at the start of week 4. Safety and tolerability assessed by adverse events enquiry, heart rate and blood pressure, 12-lead ECG, haematology and biochemistry. Efficacy assessments include Abnormal Involuntary Movement Scale (AIMS), Unified Parkinson's Disease rating Scale (UPDRS) patient PD symptom diaries, Hospital Anxiety Depression Scale (HADS), patient and clinician global impression of change in PD and dyskinesia (PGIC and CGIC).

ELIGIBILITY:
Inclusion Criteria:

* outpatient with idiopathic PD according to the UK Parkinson's Disease Society Brain Bank Clinical Diagnosis Criteria (UKPDSBBCDC)
* experiences moderately disabling dyskinesia (screening visit UPDRS 33 score≥2)
* has an mAIMS score at baseline ≥ 7 with a score ≥ 3 in at least one body area

Exclusion Criteria:

* surgical treatment for Parkinson's disease (e.g. Deep Brain Stimulation, within the last year or planned during the study)
* unstable co-existing psychiatric disease including cognitive impairment that, according to the Investigator, could interfere with the conduct of the study
* has a history of a significant medical condition that may affect the safety of the patient or preclude adequate participation in the study.
* is pregnant or breast-feeding. Female patients who are of child-bearing potential must be using adequate contraceptive methods (e.g. oral contraceptive, double-barrier method, intra-uterine device, intra-muscular hormonal contraceptive), and have a negative pregnancy test at Screening

Other protocol-defined inclusion and exclusion criteria may apply

Ages: 30 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 83 (Actual)
Dates: Start 2011-04; Primary Completion 2012-02 (Actual); Study Completion 2012-02 (Actual)

PRIMARY OUTCOMES:
Number of patients with abnormal safety and tolerability assessment parameters | 4 weeks
  Physical and neurological examination, heart rate and blood pressure, 12-lead ECG, hematology and biochemistry assessments, use of concomitant medications, adverse events and serious adverse events.

SECONDARY OUTCOMES:
Dyskinesia severity score measured by mAIMS | 4 weeks
Change in Parkinson's disease severity | 4 weeks
  Patient diary at weeks 1, 2, 3 and 4, UPDRS Part III at weeks 2 and 4, UPDRS total score at week 4
Patient-rated and clinician-rated global impression of change in dyskinesia and Parkinson's disease | 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Addex Pharma, Study Director — Addex Pharma
Locations (25):
- United States (13):
  - Addex Investigator Site, Birmingham, Alabama
  - Addex Investigator Site, Phoenix, Arizona
  - Addex Investigator Site, La Jolla, California
  - Addex Investigator Site, Los Angeles, California
  - Addex Investigator Site, Sunnyvale, California
  - Addex Investigator Site, New Haven, Connecticut
  - Addex Investigator Site, Boca Raton, Florida
  - Addex Investigator Site, Tampa, Florida
  - Addex Investigator Site, Chicago, Illinois
  - Addex Investigator Site, Southfield, Michigan
  - Addex Investigator Site, Commack, New York
  - Addex Investigator Site, Portland, Oregon
  - Addex Investigator Site, Kirkland, Washington
- Addex Investigator Site, Innsbruck, Austria
- France (5):
  - Addex Investigator Site, Bordeaux
  - Addex Investigator Site, Clermont-Ferrand
  - Addex Investigator Site, Nantes
  - Addex Investigator Site, Paris
  - Addex Investigator Site, Toulouse
- Germany (6):
  - Addex Investigator Site, Bochum
  - Addex Investigator Site, Hanau
  - Addex Investigator Site, Hanover
  - Addex Investigator Site, Kassel
  - Addex Investigator Site, Marburg
  - Addex Investigator Site, Munich

REFERENCES:
- [Derived] McFarthing K, Prakash N, Simuni T. CLINICAL TRIAL HIGHLIGHTS - DYSKINESIA. J Parkinsons Dis. 2019;9(3):449-465. doi: 10.3233/JPD-199002. No abstract available. PMID 31356217